CLINICAL TRIAL: NCT04622228
Title: Phase II, Single-Arm Study of Low-Dose Radiotherapy (LDRT) Concurrent Cisplatin/Carboplatin Plus Etoposide With Atezolizumab for Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: Study of Low-Dose Radiotherapy (LDRT) Concurrent Cisplatin/Carboplatin Plus Etoposide With Atezolizumab for Patients With Extensive-Stage Small Cell Lung Cancer
Acronym: Match
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML42391
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Small Cell Lung
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDRT concurrent cisplatin/carboplatin + etoposide + atezolizumab (Experimental): Participants will receive the following treatment regimens: LDRT concurrent cisplatin/carboplatin + etoposide + atezolizumab. Induction treatment will be administered on a 21-day cycle for four cycles. Concurrent radiation therapy will be conducted from Day 1 - Day 5 in the first cycle. Following the induction phase, participants will continue maintenance therapy with atezolizumab. Participants will be treated until loss of clinical benefit, or unaccepted toxicity, or withdrawal of consent, or death (whichever occurs first).
  Interventions: Drug: Atezolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Etoposide; Radiation: Thoracic radiation therapy (TRT)

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by intravenous infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, and clinical status.
  Other Names: Tecentriq
Drug: Cisplatin — Cisplatin will be administered as intravenous infusion at a dose of 75 mg per meter squared (75 mg/m^2) after completion of atezolizumab on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4).
Drug: Carboplatin — Carboplatin will be administered as intravenous infusion at a dose of area under the concentration-time curve (AUC) of 5 mg/mL/min on Day 1 of each 21-day cycle during the induction phase (Cycles 1-4).
Drug: Etoposide — Etoposide will be administered intravenously at a dose of 100 mg/m^2 on Days 1, 2 and 3 of each 21-day cycle during the induction phase (Cycles 1-4).
Radiation: Thoracic radiation therapy (TRT) — Participants will receive concurrent thoracic radiation therapy (TRT) treatment, in once daily fractions, 3 Gy per fraction, to a target dose of 15 Gy in 5 fractions from Day 1-Day 5 in the first cycle.

SUMMARY:
This is a Phase II, single arm, multicenter study designed to evaluate the safety and efficacy of low-dose radiotherapy (LDRT) concurrent cisplatin/carboplatin plus etoposide with atezolizumab in participants who have extensive-stage small cell lung cancer (ES-SCLC) and are chemotherapy-navïe for their extensive-stage disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ES-SCLC
* No prior treatment for ES-SCLC
* Measurable disease, as defined by RECIST v1.1. Previously irradiated lesions can be considered as measurable disease only if progressive disease has been unequivocally documented at that site since radiation.
* ECOG performance status of 0 or 1
* Life expectancy >= 3 months
* Adequate hematologic and end-organ function
* For participants receiving therapeutic anticoagulation: stable anticoagulant regimen
* Negative human immunodeficiency virus (HIV) test at screening
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following: Negative total hepatitis B core antibody (HBcAb), or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test. The HBV DNA test must be performed for participants who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test.
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening. The HCV RNA test must be performed for participants who have a positive HCV antibody test.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis
* Significant cardiovascular disease within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* History of malignancy other than small cell lung cancer (SCLC) within 5 years prior to initiation of study treatment, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | Baseline up to approximately 36 months
  Objective response rate (ORR), defined as the proportion of participants with a complete response (CR) or partial response (PR) on two consecutive occasions >= 4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Duration of Response | Baseline to disease progression or death from any cause (whichever occurs first)(up to approximately 36 months)
  Duration of response (DOR), defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Disease Control Rate (DCR) | Baseline up to approximately 36 months
  Disease control rate (DCR), defined as the proportion of participants who have a best overall response of CR or PR or stable disease (SD), as determined by the investigator according to RECIST v1.1.
Progression Free Survival (PFS) | Baseline to the first occurrence of disease progression or death from any cause (whichever occurs first) (up to approximately 36 months)
  Progression Free Survival (PFS), defined as the time from initiation of study treatment to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
PFS Rate at 6 Months and 1 Year | Baseline up to 1 year
  PFS rate at 6 months and 1 year, defined as the proportion of patients who have not experienced disease progression or death from any cause at 6 months and 1 year separately, as determined by the investigator according to RECIST v1.1.
Overall Survival (OS) | Baseline until death (up to approximately 36 months)
  OS, defined as the time from initiation of study treatment to death from any cause.
OS Rate at 1 Year and 2 Years | Baseline to 2 years or death, whichever occurs first.
  OS rate at 1 year and 2 years, defined as the proportion of patients who have not experienced death from any cause at 1 year and 2 years.
Percentage of Participants With Adverse Event | Baseline up to approximately 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- China (8):
  - Cancer Hospital , Chinese Academy of Medical, Beijing
  - Hunan Cancer Hospital, Changsha
  - West China Hospital - Sichuan University, Chengdu
  - Second Affiliated Hospital of Third Military Medical University, Chongqing
  - Shanghai Pulmonary Hospital, Shanghai
  - Fudan University Shanghai Cancer Center; Medical Oncology, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Central South Hospital, Wuhan University, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here ( https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).